CLINICAL TRIAL: NCT01485939
Title: Lidocaine Patch for Postoperative Analgesia After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Laparo_cholecystectomy_lidotop
Record Dates: First submitted 2011-11-28; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Postoperative, Pain
Keywords: lidocaine patch; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- placebo patch (Placebo Comparator)
  Interventions: Other: placebo patch applied
- lidocaine patch (Active Comparator)
  Interventions: Other: 5% lidocaine patch

INTERVENTIONS:
Other: placebo patch applied — Patients in this group would applied the placebo patch after laparoscopic cholecystectomy.
  Arms: placebo patch
Other: 5% lidocaine patch — Patients in this group would applied the 5% lidocaine patch after laparoscopic cholecystectomy.
  Arms: lidocaine patch

SUMMARY:
The investigators hypothesized that application of a 5% lidocaine patch would be associated with reduced pain scores after operation compared with placebo patch in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
* The 5% lidocaine patch have been approved for the treatment of postherpetic neuralgia.
* The investigators hypothesized that application of a 5% lidocaine patch would be associated with reduced pain scores, pain controlled drug(opioids, NSAID) in post operative period.

ELIGIBILITY:
Inclusion Criteria:

* patients of ASA Ⅰ-Ⅱ
* aged 18~65
* scheduled to undergo elective laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* patients with chronic pain
* patients with taking regular analgesics
* patients with allergy to ketorolac or lidocaine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
post operative pain after laparoscopic cholecystectomy | post operative periods
  We will measure intensity of pain(numeric rating scale)at post operative 30 minutes, 1, 2, 4, 6, 12, 24, 48 hours.

SECONDARY OUTCOMES:
pain controlled drug doses in postoperative periods. | postoperative periods
  We will measure doses of pain controlled drug(opioid, NSAIDS) at post operative 30 minutes, 1, 2, 4, 6, 12, 24, 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university Bundang hospital, Seongnam, Kyoung-ki-do, South Korea